CLINICAL TRIAL: NCT03986385
Title: Prospective, Randomized, Controlled, Multicenter, Phase III Study of Apatinib Plus Concurrent Neoadjuvant Chemoradiotherapy for Siewert II ，III of Locally Advanced HER-2 Negative Adenocarcinoma at Gastroesophageal Junction
Brief Title: Apatinib Plus Concurrent Neoadjuvant Chemoradiotherapy for Gastroesophageal Junction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Qun Zhao, Surgical director, Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRA-G04
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — XELOX

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A(apatinib Xelox) (Experimental): Preoperative: apatinib 250mg qd po q4w Capecitabine 1000mg/m2 bid d1-14，Oxaliplatin 130 mg/m2 Ivgtt d1 q3w Radiotherapy：45Gy/25f （1.8Gy/f/d，5 f/w） Postoperative: Capecitabine 1000mg/m2 bid d1-14 q3w 2 cycles
  Interventions: Drug: Apatinib Capecitabine Oxaliplatin
- B(Xelox) (Active Comparator): Preoperative: Capecitabine 1000mg/m2 bid d1-14，Oxaliplatin 130 mg/m2 Ivgtt d1 q3w Radiotherapy：45Gy/25f （1.8Gy/f/d，5 f/w） Postoperative: Capecitabine 1000mg/m2 bid d1-14 q3w 6 cycles
  Interventions: Drug: Capecitabine Oxaliplatin

INTERVENTIONS:
Drug: Apatinib Capecitabine Oxaliplatin — apatinib 250mg qd po q4w Capecitabine 1000mg/m2 bid d1-14，Oxaliplatin 130 mg/m2 Ivgtt d1 q3w
  Arms: A(apatinib Xelox)
Drug: Capecitabine Oxaliplatin — Preoperative: Capecitabine 1000mg/m2 bid d1-14，Oxaliplatin 130 mg/m2 Ivgtt d1 q3w
  Arms: B(Xelox)

SUMMARY:
The purpose of this study is to assess the efficacy and safety of patients who receive concurrent neoadjuvant chemoradiotherapy for Siewert II ，III of locally advanced HER-2 negative adenocarcinoma at gastroesophageal junction.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18 to 70 years old) at the time of voluntarily signing informed consent;
2. Histologically or cytologically confirmed adenocarcinoma. The her-2 negative was detected by immunohistochemistry or fluorescence in situ hybridization;
3. Conﬁrmed to Siewert II , III of locally advanced adenocarcinoma at gastroesophageal junction and tumor long diameter ≤8 cm by gastroscopy;
4. Patients with Stage for Ⅲ by CT/MRI (According to the eighth edition of AJCC );
5. Patients with measurable lesions(measuring≥10mm on spiral CT scan, satisfying the criteria in RECIST1.1);
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
7. Life expectancy greater than or equal to 6 months;
8. Subject must meet all of the following criteria based on the laboratory tests within 14 days prior to the first dose of study treatment.

(1) Baseline blood indicators meet the following criteria:HB≥80g/L;ANC≥1.5×109/L;PLT≥90×109/L;WBC≥4.0×109/L and ≤15×109/L (2) Baseline biochemical indicators meet the following criteria: ALT and AST≤2.5ULN, but<≤5ULN if the transferanse elevation is due to liver metastases; ALP≤2.5ULN;TBiL≤1.5ULN；Cr≤1.5ULN,Endogenous creatinine clearance rate ˃60 ml/min (Cockcroft-Gault formula);APTT≤1.5ULN,and INR or PT≤1.5ULN.

9.Women of childbearing age must have contraceptive measures or have test pregnancy (serum or urine) enroll the study before 7 days, and the results must be negative, and take the methods of contraception during the test and the last to have drugs after 8 weeks. Men must be contraception or has sterilization surgery during the test and the last to have drugs after 8 weeks; 10.Participants were willing to join in this study, and written informed consent, good adherence, cooperate with the follow-up.

Exclusion Criteria:

1. Allergic to apatinib, capecitabine and oxaliplatin;
2. The cytological examination of the abdominal cavity washing fluid showed that the tumor shedding cells were positive;
3. Have high blood pressure and antihypertensive drug treatment can not control (systolic blood pressure > 140 mmHg,diastolic blood pressure > 90 mmHg),Uncontrolled coronary heart disease and arrhythmia,classⅢ-Ⅳcardiac insufficiency;
4. A variety of factors influencing oral drugs (such as unable to swallow, nausea,vomiting,chronic diarrhea and intestinal obstruction, etc);
5. Patients with tendency of gastrointestinal bleeding, including the following:a local active ulcerative lesions,and defecate occult blood;Has melena and hematemesis in two months;
6. Coagulant function abnormality (INR > 1.5 ULN, APTT > 1.5 ULN), with bleeding tendency;
7. Pregnant or lactating women;
8. Patients with other malignant tumors within 5 years (except for curable skin basal cell carcinoma and cervical carcinoma in situ);
9. History of psychiatric drugs abuse and can't quit or patients with mental disorders;
10. Less than 4 weeks from the last clinical trial;
11. The researchers think inappropriate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
The pathological complete response rate(pCR) | [ Time Frame: within 3 weeks after surgery ]
  The lesion disappeared completely by pathology
Disease-free survival(DFS) | [ Time Frame: 3 year ]
  Baseline to measured date of recurrence or death from any cause

SECONDARY OUTCOMES:
Objective response rate (ORR) | [ Time Frame: Preoperative ]
  Baseline to measured stable disease
Disease Control Rate（DCR） | [ Time Frame: Preoperative ]
  Baseline to measured disease progression
R0-resection rate | [ Time Frame: within 3 weeks after surgery ]
  There was no residual by the microscope
Overall survival (OS) | [ Time Frame: 3years ]
  Baseline to measured date of death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- QunZhao, Shijiazhuang, Hebei, China